CLINICAL TRIAL: NCT04444687
Title: Is SARS-CoV-2 Contaminating Surgical Aerosols From Laparoscopy and Open Abdominal Surgery?
Brief Title: COVID 19: Is SARS-CoV-2 Contaminating Surgical Aerosols From Laparoscopy and Open Abdominal Surgery?
Acronym: LapCoVIDSurg
Status: Withdrawn | Type: Observational
Why Stopped: No patients
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 052020
Record Dates: First submitted 2020-06-15; First posted 2020-06-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tracheal aspirate, blood sample, fluid sample/smears from abdominal cavity, Sample from laparoscopic smoke filters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SARS-CoV-2-positive 01: SARS-CoV-2-positive patient, no symptoms, low viral load in tracheal aspirate, RNAemia not detectable
  Interventions: Diagnostic Test: Test for SARS-CoV-2
- SARS-CoV-2-positive 02: SARS-CoV-2-positive patient, symptoms, high viral load in tracheal aspirate, RNAemia not detectable
  Interventions: Diagnostic Test: Test for SARS-CoV-2
- SARS-CoV-2-positive 03: SARS-CoV-2-positive patient, symptoms, high viral load in tracheal aspirate, RNAemia detectable
  Interventions: Diagnostic Test: Test for SARS-CoV-2
- Control: Control patients, SARS-CoV-2-negative
  Interventions: Diagnostic Test: Test for SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Test for SARS-CoV-2 — * As part of normal emergency evaluation due to symptoms or following standard operation procedure for patients heading to the operating theatre the status for SARS-CoV-2 is evaluated (gene expert, Roche)
  * After intubation samples are acquired in the OR
    1. tracheal aspirate specimen directly after intubation (as part of standard operation procedures for CoVID-19 patients)
    2. blood sample (as part of standard operation procedures for CoVID-19 patients)
    3. fluid sample and smears from abdominal cavity as soon as this is accessed either by laparoscopy or laparotomy
    4. Sample from laparoscopic smoke filters (Laparoshield™ Laparoscopic Smoke Filtration System)
  * Fluid samples and smears are frozen at -80 degrees celcius for conservation in the OR.

SUMMARY:
This study aims at answering the question if aerosols from laparoscopic or open abdominal surgery contain SARS-CoV-2 virus and need to be considered contagious.

DETAILED DESCRIPTION:
The CoVID-19 pandemic has led to wide spread shut down of surgical services and restrictions to emergency procedures in most European countries and the United States. Next to concerns about resource limitations this has been justified by the risk of viral transmission during surgery. As to date the virus has been isolated from several body fluids with highest viral loads in the respiratory tract but also in feces. Aerosol producing interventions such as intubation have been proven to be a common source of health care worker infections in Italy and recently in the United Kingdom and the United States. The risk of surgical smoke and steam in open and laparoscopic surgery has been considered to bear similar risk but no data concerning these aerosols has been published so far and to the knowledge of the investigators no trials are under way (www.clinicaltrials.gov 5.4.2020). Only limited data has been available for other viral infections such as Hepatitis B and Human Papilloma Virus showing that surgical aerosols have the potential to carry such infectious particles. This rational has led to conflicting recommendations by surgical societies such as the Royal College of Surgeons or the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) to avoid laparoscopic procedures or use special filtration systems to evacuate the smoke and aerosols from the body cavity.

Since Switzerland and the city of Basel in particular currently have a high prevalence for CoVID 19 it is likely that surgeons will encounter patients with proven or suspected infection in the near future that require open or laparoscopic emergency surgical procedures. This offers the opportunity to collect a reasonable number of samples and smears from the abdominal cavity and surgical aerosols from these patients in limited time to answer the urgent question whether surgical smoke and aerosols of the abdominal cavity from CoVID-19 patients are contagious or not.

Investigators consider the trial to be a risk category A according to art 7 (HRO). There is no risk for patients included in this trial since the treatment of the patients will not differ from standard care. There will be no extra tests performed and only routine data will be collected. Specimen from laparoscopic smoke filters which are a protection device for medical staff will be tested on SARS-CoV-2 contamination.

Primary Objective:

The primary objective of the study is to investigate the contamination of surgical smoke and aerosols with SARS-COV-2 virus particles using the viral genome as a marker during laparoscopic and open abdominal emergency procedures for patients with suspected or proven infection.

Secondary objectives are to:

* assess the viral load in the peritoneal cavity and fluid
* compare viral load of smoke and aerosols in laparoscopic and open procedures
* assess possible transmission to surgeons during their service

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Proven or suspected (not ruled out) SARS-CoV-2 infection (at the time of surgery)
* Undergoing urgent or emergency laparoscopic or open abdominal surgery
* Able to provide informed general consent on further use of clinical data

Exclusion Criteria:

* Age < 18 years
* Unable to provide informed general consent & no possibility of informed general consent by proxy
* Recent (<24h) negative test for SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inhabitants of the area around Basel/North west Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
SARS-COV-2 RNA detection | Up to 12 months
  The primary outcome will be SARS-COV-2 RNA detection in filter systems for surgical aerosols in laparoscopic surgery (YES/NO).
  If viral RNA can be detected, the aerosols should be considered contagious, and therefore the debate on protective measures for the surgical staff in case of emergency surgery and possibly delaying any urgent surgery to protect surgical teams would be reasonable.
  If viral RNA cannot be detected, the aerosols do not need to be considered contagious for SARS-CoV-2, and CoVID-19 patients could safely be considered for laparoscopic and open abdominal surgery if indicated.

SECONDARY OUTCOMES:
Viral contamination of peritoneal cavity and fluid | Up to 12 months
  Viral contamination of peritoneal cavity and fluid in laparoscopic cases (YES/NO)
Viral contamination of peritoneal cavity and fluid in open cases | Up to 12 months
  Viral contamination of peritoneal cavity and fluid in open cases (YES/NO)
Viral infection of members of the surgical team | Up to 12 months
  Viral infection of members of the surgical team (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Marco von Strauss und Torney, Principal Investigator — Clarunis University Centre for Gastrointestinal and Liver Diseases

IPD SHARING:
Plan to Share IPD: No